CLINICAL TRIAL: NCT00014625
Title: Open Label Phase II Study Of E7070 In Patients With Metastatic Melanoma (Stage IV)
Brief Title: E7070 in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16005-18002; EORTC-16005; EORTC-18002; EISAI-E7070-E044-205
Record Dates: First submitted 2001-04-10; First posted 2004-02-16 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — N-(3-chloro-7-indolyl)-1,4-benzenedisulphonamide

INTERVENTIONS:
Drug: indisulam

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of E7070 in treating patients who have stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the therapeutic activity of E7070 in terms of objective response, duration of response, and progression-free survival of patients with metastatic melanoma. II. Determine the acute side effects of this drug in these patients. III. Determine the pharmacokinetic parameters of this drug in these patients.

OUTLINE: This is a multicenter study. Patients receive E7070 IV over 1 hour. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed every 6 weeks.

PROJECTED ACCRUAL: A total of 19-24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage IV melanoma Metastatic disease At least 1 bidimensionally measurable target lesion by CT scan No brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 OR WHO 0-2 Life expectancy: Not specified Hematopoietic: Hemoglobin greater than 10 g/dL Neutrophil count greater than 2,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 2.5 times ULN (5 times ULN if liver metastases present) Transaminases no greater than 2.5 times ULN (5 times ULN if liver metastases present) Renal: Creatinine no greater than 1.7 mg/dL Cardiovascular: Clinically normal cardiac function No history of severe or unstable ischemic heart disease 12-lead ECG normal Other: No history of unstable systemic disease No concurrent uncontrolled diabetes mellitus No concurrent infection No history of hypersensitivity to sulfonamides No other malignancy within the past 5 years except cone-biopsied carcinoma of the cervix or adequately treated basal cell or squamous cell skin cancer No psychological, familial, sociological, or geographical condition that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 2 weeks since prior blood transfusions At least 2 weeks since prior growth factors At least 6 weeks since prior experimental vaccine therapy No prior immunotherapy for metastatic disease No concurrent anticancer immunotherapy Chemotherapy: No prior chemotherapy for metastatic disease No other concurrent anticancer chemotherapy Endocrine therapy: No concurrent anticancer hormonal therapy Radiotherapy: No concurrent anticancer radiotherapy except palliation for pain control or other reasons (e.g., bronchial obstruction or ulcerating skin lesions) with no curative intent Surgery: Not specified Other: At least 6 weeks since prior adjuvant or neoadjuvant therapy At least 4 weeks since prior experimental drugs At least 2 weeks since prior and no concurrent coumarin anti-coagulants, terfenadine, cisapride, cyclosporine, tacrolimus, theophylline, diazepam, sulfonylurea anti-diabetics, phenytoin, or carbamazepine No other concurrent experimental agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2001-02; Primary Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F. Smyth, MD, Study Chair — Edinburgh Cancer Centre at Western General Hospital; Steinar Aamdal, MD, PhD, Study Chair — Norwegian Radium Hospital
Locations (12):
- Kaiser Franz Josef Hospital, Vienna, Austria
- Institut Jules Bordet, Brussels, Belgium
- France (3):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - Centre Eugene Marquis, Rennes
- Medizinische Hochschule Hannover, Hanover, Germany
- Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples, Italy
- Norwegian Radium Hospital, Oslo, Norway
- Instituto Portugues de Oncologia de Francisco Gentil, Lisbon, Portugal
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- United Kingdom (2):
  - Royal Marsden NHS Trust, London, England
  - Western General Hospital, Edinburgh, Scotland

REFERENCES:
- [Result] Smyth JF, Aamdal S, Awada A, Dittrich C, Caponigro F, Schoffski P, Gore M, Lesimple T, Djurasinovic N, Baron B, Ravic M, Fumoleau P, Punt CJ; EORTC New Drug Development and Melanoma Groups. Phase II study of E7070 in patients with metastatic melanoma. Ann Oncol. 2005 Jan;16(1):158-61. doi: 10.1093/annonc/mdi016. PMID 15598954